CLINICAL TRIAL: NCT05678166
Title: Validation of Soluble Programmed Death-1 in Predicting Progression of Nodular-bronchiectatic Form of Nontuberculous Mycobacterial Lung Disease: a Multi-Country Research
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202210007RINC
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-09

CONDITIONS: Nontuberculous Mycobacterial Lung Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NTM-LD: Diagnosis is made on the basis of the guidelines produced by the American Thoracic Society . Briefly, Patients have pulmonary symptoms with identified chest image and fit with the microbiology criteria.
- NTM pulmonary colonizers and others: Those without fulfilling the diagnostic criteria but having at least one set of positive sputum for MAC or patients infected with NTM other than MAC species.
- Pulmonary tuberculosis (TB): Those with respiratory specimen culture positive for Mycobacterium tuberculosis or typical TB pulmonary pathology.
- Healthy control: Healthy control

SUMMARY:
The incidence of nontuberculous mycobacterial lung disease (NTM-LD) is increasing worldwide and in Eastern Asia. NTM-LD leads significant morbidity and mortality, around 25% within 5 years, but the treatment rate is low because the course of NTM-LD is indolent, especially in nodular-bronchiectatic (NB) form. However, there is no biomarker proven for predicting the progression in NB form of NTM-LD. Recently, it has been reported that the ratio of membrane-form programmed death-1 (PD-1) expressed T cells increased in patients with NTM-LD and it was associated with disease severity and progression. The mechanism has been speculated as a "immune exhaustion". In contrast to PD-1 expressed in cell membrane, soluble-form PD-1 is another biomarker that can be easily detected in serum. We recently reported that soluble PD-1 significantly correlated with cavitary lesion and disease progression in patients with NB-form NTM-LD in Taiwan. However, this has not been validated in other countries and ethnicities. Furthermore, the usefulness of soluble PD-1 in diagnosis and predicting mortality warrants further studies.

DETAILED DESCRIPTION:
The incidence of nontuberculous mycobacterial lung disease (NTM-LD) is increasing worldwide and in Eastern Asia. NTM-LD leads significant morbidity and mortality, around 25% within 5 years, but the treatment rate is low because the course of NTM-LD is indolent, especially in nodular-bronchiectatic (NB) form. However, there is no biomarker proven for predicting the progression in NB form of NTM-LD. Recently, it has been reported that the ratio of membrane-form programmed death-1 (PD-1) expressed T cells increased in patients with NTM-LD and it was associated with disease severity and progression. The mechanism has been speculated as a "immune exhaustion". In contrast to PD-1 expressed in cell membrane, soluble-form PD-1 is another biomarker that can be easily detected in serum. We recently reported that soluble PD-1 significantly correlated with cavitary lesion and disease progression in patients with NB-form NTM-LD in Taiwan. However, this has not been validated in other countries and ethnicities. Furthermore, the usefulness of soluble PD-1 in diagnosis and predicting mortality warrants further studies. Moreover, it is worthwhile to measure soluble PD-1 in bronchoalveolar lavage to explore local immune pathogenesis of NTM-LD. Therefore, we apply this project to investigate the role of soluble PD-1 in NTM-LD through a multi-country cooperation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* NTM-LD: (N=250) Diagnosis is made on the basis of the guidelines produced by the American Thoracic Society.Patients have pulmonary symptoms with identified chest image and fit with the microbiology criteria.
* NTM pulmonary colonizers and others: (N=100) Those without fulfilling the diagnostic criteria but having at least one set of positive sputum for MAC or patients infected with NTM other than MAC species.
* Pulmonary tuberculosis (TB): (N=100) Those with respiratory specimen culture positive for Mycobacterium tuberculosis or typical TB pulmonary pathology.
* Healthy control (N=50)

Exclusion Criteria:

* Patients who have acquired immunodeficiency syndrome

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with NTM-LD at National University Hospital, Taiwan ,Fukujuji Hospital, Japan and Seoul National University, Korea.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-31 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma soluble PD-1 on NTM-LD diagnosis | within 2 years
Mortality | within 2 years
  Mortality, patient die within 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan